CLINICAL TRIAL: NCT00523367
Title: COPD Patients Diagnosed With Gastro Esophageal Reflux Disease Have Decreased Rates of COPD Exacerbations After Treatment With High Dose Proton Pump Inhibitor Therapy (Esomeprazole or Lansoprazole)
Brief Title: COPD Patients Diagnosed With GERD,COPD Exacerbations After Treatment With High Dose PPI
Acronym: GERD/COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated due to enrollment
Sponsor: University of Florida (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-L-147
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2012-07-24 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Gastroesophageal Reflux; Chronic Obstructive Pulmonary Disease
Keywords: Gastro Esophageal Reflux Disease (GERD); Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Gastroesophageal Reflux; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- esomeprazole (No Intervention)
  Interventions: Procedure: 24 hour pH testing

INTERVENTIONS:
Procedure: 24 hour pH testing — 24 hour pH testing will be used to screen patients
  Other Names: Pevacid

SUMMARY:
The purpose of this study is to determine which COPD patients have GERD and if COPD patients with GERD treated with high dose lansoprazole for 1 year decreases the frequency of COPD exacerbations compared to the previous year without treatment.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a common esophageal disorder with 40% of the US adult population experiencing symptoms monthly. Pulmonary diseases associated with GERD may include pneumonia, pulmonary fibrosis, asthma, or chronic bronchitis. The latter may be a manifestation of chronic obstructive pulmonary disease (COPD), suggesting GERD as a risk factor for acute exacerbation of COPD. Acute exacerbations of COPD are a major cause of morbidity and mortality in patients with the disease. Recent work suggests that COPD patients with a minimum of weekly reflux symptoms have an increased number of COPD exacerbations that those who are either asymptomatic or have GERD symptoms less than once a week. On this basis, we theorized that in patients with COPD, who also have gastro esophageal reflux disease are at increase risk for acute exacerbations of COPD. To test this question, we will determine which COPD patients have GERD by 24 hour pH testing, treat their GERD with esomeprazole or lansoprazole for 1 year, and compare the number of COPD exacerbations during the treatment period to the previous year.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD
* forced expiratory volume/forced vital capacity ratio (FEV1/FVC) of < 70% on pulmonary function testing
* age > 40 years
* >20 pack year history of smoking

Exclusion Criteria:

* presence of the following disorders: respiratory disorders other than COPD, known esophageal disease such as cancer, achalasia, stricture, active peptic ulcer disease, Zollinger-Ellison syndrome, mastocytosis, scleroderma, or current abuse of alcohol defined as greater than three alcoholic drinks per day.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Munoz, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: University of Florida Research Studies — http://www.hscj.ufl.edu/medicine/research-affairs/search/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A flyer was posted in the pulmonary clinic which provides basic information about the trial and instructs the reader to ask their doctor for more information. Interested patients were referred to the Gastroenterology Clinic where they were consented and screened.
Pre-assignment Details: Eligible patients with a known diagnosis of COPD and pulmonary function testing meeting criteria were asked to complete a validated GERD and quality of life questionnaire. These questionnaires are queried for GERD symptoms and an assessment of overall health during the previous year.
Groups:
- COPD Patients With GERD Symptoms: Patients with a diagnosis of COPD with weekly GERD symptoms will be asked to complete GERD and quality of life questionnaires. These questionnaires queried for GERD symptoms and an assessment of overall health during the previous year.
Period: Overall Study
Arm/Group | COPD Patients With GERD Symptoms
Started | 25
Completed | 2
Not Completed | 23
Not completed — 19 screen failures | 19
Not completed — 4 Withdrawn by PI | 4

BASELINE CHARACTERISTICS:
Arm/Group | COPD Patients With GERD Symptoms
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 59.16 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gastro Esophageal Reflux Disease One Year After Treatment.
Description: The number of participants who have Gastro Esophageal Reflux Disease after one year of treatment.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | COPD Patients With GERD Symptoms
Number analyzed (Participants) | 2
participants | 0

2. Secondary Outcome: COPD/GERD Patients Treated With High Dose Esomeprazole
Description: COPD patients with GERD treated with high dose esomeprazole for 1 year decreases the frequency of COPD exacerbations compared to the previous year without treatment.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | COPD Patients With GERD Symptoms
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 4/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPD Patients With GERD Symptoms (N=25)
Cough (General disorders) | 1 (1)
Shortness of breath (General disorders) | 1 (1)
Sore throat (General disorders) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2)
Nausea (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Increased COPD (General disorders) | 2 (2)
Flu symptoms (General disorders) | 1 (1)
Hemoptysis (General disorders) | 1 (1)
Bronchitis (General disorders) | 1 (2)
Dizziness (General disorders) | 1 (1)
Sinusitis (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No